CLINICAL TRIAL: NCT00989976
Title: Individual Differences in Diabetes Risk: Role of Sleep Disturbances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: #16028A; DOD PR064727
Record Dates: First submitted 2009-10-01; First posted 2009-10-06 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Sleep; Diabetes
Keywords: Sleep; Diabetes Risk
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 8.5 h sleep (Other): Subjects will have normal sleep times
  Interventions: Behavioral: normal sleep times
- restricted bedtimes (Other): 4.5 h bedtimes
  Interventions: Behavioral: bedtime restriction

INTERVENTIONS:
Behavioral: normal sleep times — 8.5 h bedtimes
  Arms: 8.5 h sleep
Behavioral: bedtime restriction — 4.5 h restricted bedtimes
  Arms: restricted bedtimes

SUMMARY:
The hypothesis for this study is that some individuals may be at much higher risk to develop type 2 diabetes and that the individual diabetes risk will be predicted by the individual level of slow wave sleep activity (SWA).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women with low Slow Wave Sleep Activity (SWA) or high SWA with the gender distribution in each group matching the gender distribution of active duty Army personnel (85% men; 15% women) based on the following inclusion criteria:

  * age 18 to 29 years,
  * normal weight or modestly overweight (BMI ≤ 27 kg/m2 for women, BMI ≤ 28 kg/m2 for men),
  * normal findings on clinical examination, normal routine laboratory tests results, normal EKG, no history of psychiatric, endocrine, cardiac or sleep disorders.
* Only subjects who have regular life styles (no shift work, no travel across time zone during the past 4 weeks), habitual bedtimes between 7.0-8.5 hours, and do not take medications will be recruited.
* An overnight polysomnography will be performed to rule out sleep-disordered breathing (apnea-hypopnea index > 5/hour) and periodic limb movement disorder (PLM arousal index >1/hour).
* Women taking hormonal contraceptive therapy and pregnant women will be excluded. In women, all studies will be initiated in the early follicular phase.

Exclusion Criteria:

* Tobacco use.
* Habitual alcohol use of more than 2 1 drink per day.
* Excessive caffeine intake of more than 300 mg per day and individuals with a metal implant or another metal object in their body.

We estimate that we will need to recruit at least 60-70 individuals to obtain two gender-matched groups of 16 individuals with either low or high SWA.

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
diabetes risk as assessed by disposition index | Dec. 2011

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, PhD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States